CLINICAL TRIAL: NCT07176000
Title: Strengthening Awareness and Community Resources for Early Detection of Lung Cancer Through Navigation Guided Screening Trial (SACRED LUNGS Aims 1.2-3)
Brief Title: Tailored Patient Navigation to Improve the Uptake of Lung Cancer Screening in Tribal Communities in Western Washington State, SACRED LUNGS Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RG1125421; NCI-2025-06016 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020813 (Other: Fred Hutch/University of Washington Cancer Consortium); U19MD020533 (NIH)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Navigation; Early Intervention, Educational; Educational Status; Methods; Practice Guidelines as Topic; Standard of Care; Interviews as Topic

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research staff and study coordinators will be blinded to study arm while patient, navigators, and providers will be aware of study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (tailored PN) (Experimental): Participants receive tailored PN activities in support of the uptake and follow-up of LCS for 21 months. Participants also receive an educational handout on LCS on study.
  Interventions: Behavioral: Patient Navigation; Other: Educational Intervention; Other: Interview; Other: Survey Administration; Other: Electronic Health Record Review
- Arm 2 (enhanced usual care, delayed tailored PN) (Active Comparator): Participants receive enhanced usual care consisting of an educational handout on LCS and a warm hand-off to discuss LCS with their PCP for 6 months. Participants then receive tailored PN services in support of the uptake and follow-up of LCS for 15 months.
  Interventions: Behavioral: Patient Navigation; Other: Best Practice; Other: Interview; Other: Survey Administration; Other: Electronic Health Record Review

INTERVENTIONS:
Behavioral: Patient Navigation — Receive tailored PN activities
  Other Names: Patient Navigator Program
Other: Educational Intervention — Receive LCS educational handout
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm 1 (tailored PN)
Other: Best Practice — Receive enhanced usual care
  Other Names: standard of care; standard therapy
  Arms: Arm 2 (enhanced usual care, delayed tailored PN)
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial studies whether tailored patient navigation (PN) works to improve the uptake of lung cancer screening (LCS) in tribal communities in western Washington state. Lung cancer is the leading cause of cancer death in the United States among American Indian (AI) and Alaska Native (AN) people, and the incidence of lung cancer is higher in this population in the Northern and Southern Plains, Alaska, and Pacific Coast regions. In Washington state, AI/AN people also have twice the rate of commercial cigarette smoking than the overall population. LCS with annual low-dose chest computed tomography (CT) can reduce lung cancer death and is recommended in people 50-80 years of age with current or recent (within 15 years) tobacco use and a 20 pack-year or greater smoking history. Despite this, AI and AN people are less likely to receive LCS which may be due to barriers they face making it difficult to receive LCS. PN services are designed to guide a patient through the healthcare system and reduce barriers to timely screening, follow-up, diagnosis, treatment, and supportive care. The PN services in this trial have been tailored for the tribal communities in western Washington state. The services are designed to help participants overcome the unique barriers that their tribal communities face and improve the uptake of LCS.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM 1: Participants receive tailored PN activities in support of the uptake and follow-up of LCS for 21 months. Participants also receive an educational handout on LCS on study.

ARM 2: Participants receive enhanced usual care consisting of an educational handout on LCS and a warm hand-off to discuss LCS with their primary care physician (PCP) for 6 months. Participants then receive tailored PN services in support of the uptake and follow-up of LCS for 15 months.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1.2 RANDOMIZED CONTROLLED TRIAL: Between ages 50-77
* AIM 1.2 RANDOMIZED CONTROLLED TRIAL: Self-reported 20-pack year smoking history
* AIM 1.2 RANDOMIZED CONTROLLED TRIAL: Ongoing commercial tobacco use within the past 15 years
* AIM 1.2 RANDOMIZED CONTROLLED TRIAL: Seen by a PCP at a participating clinic (South Puget Intertribal Planning Agency [SPIPA] or Muckleshoot) within the past three years

  * Potential participants who want to establish care at an eligible clinic will be connected to a PCP
* AIM 2 CLINICAL STAFF SURVEYS AND SEMI-STRUCTURED INTERVIEWS: At least 18 years of age
* AIM 2 CLINICAL STAFF SURVEYS AND SEMI-STRUCTURED INTERVIEWS: Affiliation with Muckleshoot or SPIPA (one of the 6 community partnering clinics) as a provider, or supportive staff member
* AIM 2 PATIENT SURVEYS AND SEMI-STRUCTURED INTERVIEWS: Patient participated in the aim 1.2 trial
* AIM 3 CLINICAL STAFF SURVEYS AND SEMI-STRUCTURED INTERVIEWS: At least 18 years of age
* AIM 3 CLINICAL STAFF SURVEYS AND SEMI-STRUCTURED INTERVIEWS: Affiliation with Muckleshoot or SPIPA (one of the 6 community partnering clinics) as a provider, or supportive staff member
* AIM 3 PATIENT SURVEYS AND SEMI-STRUCTURED INTERVIEWS: Patient participated in the aim 1.2 trial

Exclusion Criteria:

* AIM 1.2 RANDOMIZED CONTROLLED TRIAL: Has had a documented chest CT within the past one year
* AIM 1.2 RANDOMIZED CONTROLLED TRIAL: Personal history of lung cancer or symptoms associated with lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-29 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion of chest computed tomography (CT) (Aim 1.2) | Up to 6 months
  Will be compared between arms using the Cochran-Mantel-Haenszel (CMH) test, accounting for the stratification variables used during randomization. Completion rates will also be estimated in each arm and 95% confidence intervals for the rates and their difference will be calculated using Wilson's score method. The single primary outcome will be tested using two-sided α = 0.05.

SECONDARY OUTCOMES:
Completion of low dose computed tomography of the chest (Aim 1.2) | Up to 21 months
  Will be compared between arms using the CMH test. Will be tested using two-sided α = 0.05 without adjustment for multiplicity.
Lung cancer screening (LCS) knowledge (Aim 1.2) | At 21 months
  Will be compared between arms using a stratified Wilcoxon rank-sum test (van Elteren test). Will be tested using two-sided α = 0.05 without adjustment for multiplicity.
Health-related quality of life (Aim 1.2) | At 21 months
  Will be measured using the Short Form 36 Health Survey questionnaire. Will be compared between arms using a stratified Wilcoxon rank-sum test (van Elteren test). Will be tested using two-sided α = 0.05 without adjustment for multiplicity.
Rate of reported 30-day cessation period (Aim 1.2) | Up to 6 months
  The impact of navigation on tobacco cessation will be explored by the rates of a reported 30-day cessation period during the intervention period as measured by self-reported 30-day floating abstinence.
Completion of chest CT (Aim 2) | Up to 6 months
  Quantitative analyses will use structural equation models (SEM) to understand the relationships between measured and latent variables representing barriers, facilitators and social determinants of health and the outcome of CT completion.
Navigation care engagement (Aim 2) | Up to 21 months
  Quantitative analyses in this aim will use SEM to understand the relationships between measured and latent variables representing barriers, facilitators and social determinants of health and the outcome of navigation care engagement. Measure of reach will be operationalized as an ordinal scale based on care completion activities along the LCS continuum as documented in the electronic health record.
Completion of chest CT (Aim 3) | Up to 15 months
  The rate of chest CT completion during the maintenance phase in the control arm (after navigation is offered) will be estimated and compared with the rate during the trial phase (before navigation was offered) using Poisson regression with the log link. The phase (trial versus maintenance) will be modeled using a time varying covariate, where each participant will contribute an outcome for each phase in which they are still "at risk" for completing CT (i.e., until first CT completion or end of follow-up). Models will include additional key covariates, including clinical site, smoking status, and prior reported LCS. Generalized estimating equations will be used to account for multiple periods per participant and potential overdispersion.
Completion of next diagnostic step in LCS follow-up | Up to 15 months
  Adherence to follow-up will be assessed as binary completion of the next step in follow-up among those with a completed chest CT during the randomized controlled trial. Appropriate next step in follow-up is determined through the Lung CT Screening Reporting and Data System (Lung-RADS) system, with most participants having negative initial CT (Lung-RADS 1 or 2) with follow-up assessed at 11-15 months. Adherence rates will be estimated as a proportion with 95% confidence intervals, summarized overall and stratified by Lung-RADS.

CONTACTS AND LOCATIONS:
Overall Officials: Matty Triplette, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Muckleshoot Tribal Clinic, Auburn, Washington
  - South Puget Intertribal Planning Agency (SPIPA), Shelton, Washington

IPD SHARING:
Plan to Share IPD: No